CLINICAL TRIAL: NCT05962450
Title: An Open Label, Randomized, Controlled, Clinical Trial of Adoptive Autologous Invariant Natural Killer T Cells for the Treatment of Progressed Hepatocellular Carcinoma Continuing on PD-1 Inhibitor Therapy
Brief Title: Adoptive Autologous iNKT Cells for the Treatment of Progressed Hepatocellular Carcinoma Continuing on PD-1 Inhibitor Therapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing YouAn Hospital (Other)
Collaborators: Beijing Gene Key Life Technology Co., Ltd (Industry)
Responsible Party: Principal Investigator, LU JUN, Chief physician, Beijing YouAn Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Beijing YouAn Ethics [2023]060
Record Dates: First submitted 2023-07-04; First posted 2023-07-27 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — regorafenib

STUDY DESIGN:
Masking Description: Block randomization was performed by the independent masked statistician. Two independent masked radiologist who are blinded to patients' clinical information will review the imaging examinations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RPI group (Experimental): Regorafenib + PD-1 + iNKT cells
  Interventions: Biological: iNKT Cells; Drug: PD-1; Drug: Regorafenib
- RP group (Other): Regorafenib + PD-1
  Interventions: Drug: PD-1; Drug: Regorafenib

INTERVENTIONS:
Biological: iNKT Cells — the iNKT cells will be intravenous infused every two weeks as a course of treatment for up to six courses , the reinfusion dose is determined according to the patient's body surface area, which was about 108~109cells/m2.
  Other Names: Vα24+ T Cells
  Arms: RPI group
Drug: PD-1 — Intravenous infusion, according to the drug instructions.
Drug: Regorafenib — Oral administration, according to the drug instructions.

SUMMARY:
The goal of this clinical trial is to explore the efficacy and safety of autologous iNKT cells in patients with progressed hepatocellular carcinoma (HCC) after treatment with PD-1 antibody. The main question it aims to answer are:

* the efficacy of autologous iNKT cells in patients with progressed HCC after treatment with PD-1 antibody.
* the safety of autologous iNKT cells in patients with progressed HCC after treatment with PD-1 antibody.

Participants will be randomized 1:1 to receive Regorafenib + PD-1 + iNKT cells (RPI group) or the treatment of Regorafenib + PD-1 (RP group).

Researchers will compare RPI group and RP group to see whether the iNKT cells can achieve a better therapeutic effect on HCC patients with PD-1 resistance.

DETAILED DESCRIPTION:
Single center, randomized, open trial in Barcelona Clinic Liver Cancer（BCLC）C stage patients with progressed HCC after anti-angiogenic targeted drugs combined with PD-1 monoclonal antibody therapy to explore the efficacy and safety of autologous iNKT cells.

This study includes screening period, treatment period and follow-up period (until the subjects withdrew their informed consent or received other anti-tumor therapy or participated in other clinical trials or the researchers judged that it is not in the best interests of patients to continue to participate in the study) after treatment.

The patients will be randomized 1:1 using a random number table to receive Regorafenib + PD-1 + iNKT cells (RPI group) or the treatment of Regorafenib + PD-1 (RP group).

1. iNKT Cells：Intravenous infusion. The cells will be infused every two weeks as a course of treatment for up to six courses.
2. PD-1：Intravenous infusion, according to the drug instructions.
3. Regorafenib：Oral administration, according to the drug instructions. All target and non-target lesions will be assessed by chest, abdomen, and pelvis CT or MRI at baseline and every 8 weeks until radiological progression (according to mRECIST/iRECIST).

Safety and side-effect profiles will be assessed based on the nature, frequency, and severity of adverse events, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years of age.
* Barcelona Clinic Liver Cancer（BCLC） C stage hepatocellular carcinoma (HCC) confirmed by CT, MRI, and/or histopathology.
* Progressed after receiving anti-angiogenic targeted drugs combined with PD-1 monoclonal antibody.
* Life expectancy of at least 12 weeks.
* Child-Pugh A/B.
* Voluntary signing of informed consent.

Exclusion Criteria:

* History of severe hypertension or cardiac disease.
* known central nervous system (CNS) tumor or combined with other malignant disorders.
* Uncontrolled immune system or infectious disease.
* Known history of the human immunodeficiency virus (HIV) or syphilis infection.
* History of stem cell transplant or organ allograft.
* History of allergy to immunotherapy or related drugs.
* Bilirubin is twice times the upper limit of normal.
* Glomerular filtration rate （GFR）< 60ml/min.
* Serious complications include moderate or severe infective pleural and peritoneal effusion, pericardial effusion, upper gastrointestinal bleeding, hepatic encephalopathy.
* Pregnancy or lactation.
* History of severe allergy to any monoclonal antibody or anti-angiogenic targeted drug.
* Deemed not suitable for cellular immunotherapy by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | The time from enrollment to disease progression, or death from any cause, whichever occurred first, up to 24 months.
  The time from enrollment to disease progression according to the modified RECIST (mRECIST) guideline in trial immunotherapeutics, or death from any cause, whichever occurred first；the time from enrollment to confirmed disease progression (iCPD) according to the iRECIST

SECONDARY OUTCOMES:
Disease control rate (DCR) | Evaluation was performed every 8 weeks after the start of the treatment, up to 24 months.
  including complete response (CR), partial response (PR), and disease stabilization (SD), evaluated by imaging according to iRECIST for target lesions and assessed by MRI/CT.
Objective response rate (ORR) | Evaluation was performed every 8 weeks after the start of the treatment, up to 24 months.
  complete response (CR) and partial response (PR) evaluated by imaging according to mRECIST/iRECIST for target lesions and assessed by MRI/CT.
Overall survival (OS) | Time from the date of enrollment to the date of death from any cause, up to 36 months.
  Time from the date of enrollment to the date of death from any cause.
1-year overall survival rate (1-year OS rate) | Time from the date of enrollment to 1 year later.
  The proportion of subjects who were still alive from the date of enrollment to 1 year later
Duration of Overall Response (DOR) | Time from the first tumor remission to the first recording of disease progression or death from any cause, up to 24 months..
  The time from the first tumor remission (CR or PR according to mRECIST/iRECIST) to the first recording of disease progression (PD according to mRECIST criteria or iCPD according to iRECIST) or death from any cause (whichever occurs first).
Time to progression (TTP) | Time from the date of enrollment to the date of first disease progression, up to 24 months.
  Time from the date of enrollment to the date of first disease progression (PD) according to mRECIST or iCPD according to iRECIST).
Time to Quality of Life (QoL) Deterioration | Time from the date of enrollment, up to 24 months.
  EORTC QLQ-C30: European Organization for Research on Treatment of Cancer Quality of Life Questionnare-Core 30.
  The totally 30 items spread out over five functional scales (15 items), three symptom scales (7 items), a global health status/QoL scale (2 items), and six single items. 1-28 item ranges 1: not at all, 2: a little, 3: quite a lit, 4: very much; 29-30 item ranges 1-7 from very poor to excellent. Raw score (RS) is an average of all items in each area. Standardized score is in the range of 0-100 by formula SS=[1-(RS-1)/n] x100 (function) or SS=[（RS-1）/n]x100 (symptom or overall health) respectively. A high scale score represents a higher/healthy response level.
  Time to deterioration was defined as a decrease from baseline of 10 points or more on the EORTC QLQ-C30 maintained for two consecutive assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Lu, MD., Principal Investigator — Beijing YouAn Hospital
Locations (1):
- Beijing Youan Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No